CLINICAL TRIAL: NCT00695838
Title: Evaluation of the Impact of Abdominal Fat on GERD Severity and GERD Frequency in General Practice
Brief Title: National Survey on Gastroesophageal Reflux Disease (GERD) Patients
Acronym: LINEA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GFR-DUM-2007/3
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: GERD
Keywords: GERD symptoms- Waist circumference; Patients with symptomatic GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this observational study is to assess the impact of abdominal fat on severity and frequency of GERD symptoms .

ELIGIBILITY:
Inclusion Criteria:

* Male or female > or = 18 years old
* Patient with symptomatic GERD
* Without PPI or H2 antagonist treatment during the 3 previous months
* Agree to take part in this study

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First three consecutive patients with GERD symptoms seen by GP
Sampling Method: Probability Sample
Enrollment: 5084 (Actual)
Dates: Start 2008-01; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Waist circumference | Once

SECONDARY OUTCOMES:
Frequency of GERD symptoms | Once
GERD impact scale | Once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Medical Director, Study Director — AstraZeneca
Locations (1624):
- France (1624):
  - Research Site, Ablon-sur-Seine
  - Research Site, Achenheim
  - Research Site, Afa
  - Research Site, Agde
  - Research Site, Agen
  - Research Site, Agneaux
  - Research Site, Aigre
  - Research Site, Aigrefeuille SUR MAI
  - Research Site, Aire-sur-la-Lys
  - Research Site, Aiserey
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Ajaccio
  - Research Site, Alba-la-Romaine
  - Research Site, Albertville
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Ambazac
  - Research Site, Ambès
  - Research Site, Ambierle
  - Research Site, Ambilly
  - Research Site, Ambleteuse
  - Research Site, Amboise
  - Research Site, Amelie LES Bains CED
  - Research Site, Amiens
  - Research Site, Amphion-les-Bains
  - Research Site, Amplepuis
  - Research Site, Andernos-les-Bains
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Angers
  - Research Site, Anglet
  - Research Site, Angoulême
  - Research Site, Aniche
  - Research Site, Annay
  - Research Site, Annecy
  - Research Site, Annecy-le-Vieux
  - Research Site, Annezin
  - Research Site, Annonay
  - Research Site, Anse
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Anzin
  - Research Site, Apprieu
  - Research Site, Apt
  - Research Site, ARC ET Senans RC ET Senans
  - Research Site, Arcachon
  - Research Site, Arches
  - Research Site, Argences
  - Research Site, Argentat
  - Research Site, Argenteuil
  - Research Site, Argentré-du-Plessis
  - Research Site, Arles
  - Research Site, Armentières
  - Research Site, Arpajon
  - Research Site, Arradon
  - Research Site, Arras
  - Research Site, Art-sur-Meurthe
  - Research Site, Artenay
  - Research Site, Arthon-en-Retz
  - Research Site, Arudy
  - Research Site, Arzano
  - Research Site, Arzon
  - Research Site, Asnières-sur-Seine
  - Research Site, Aspiran
  - Research Site, Asson
  - Research Site, Athies
  - Research Site, Athis-Mons
  - Research Site, Aubagne
  - Research Site, Aubenas
  - Research Site, Aubervilliers
  - Research Site, Aubière
  - Research Site, Aubigny
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Auchy-les-Mines
  - Research Site, Audruicq
  - Research Site, Audun-le-Roman
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aumale
  - Research Site, Auray
  - Research Site, Aurillac
  - Research Site, Auriol
  - Research Site, Authon-du-Perche
  - Research Site, Autun
  - Research Site, Auxerre
  - Research Site, Auxonne
  - Research Site, Availles-Limouzine
  - Research Site, Avelin
  - Research Site, Avesnelles
  - Research Site, Avesnes-les-Aubert
  - Research Site, Avignon
  - Research Site, Axat
  - Research Site, Aytré
  - Research Site, Azay-le-Ferron
  - Research Site, Azerailles
  - Research Site, Badevel
  - Research Site, Bagneux Saumur
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baillargues
  - Research Site, Bailleul
  - Research Site, Balan
  - Research Site, Balbigny
  - Research Site, Ballon
  - Research Site, Balma
  - Research Site, Bapaume
  - Research Site, Bar-le-Duc
  - Research Site, Barbezieux Saint Hilair
  - Research Site, Barentin
  - Research Site, Barlin
  - Research Site, Basse-Goulaine
  - Research Site, Bassussarry
  - Research Site, Bastia
  - Research Site, Baugé
  - Research Site, Baulon
  - Research Site, Baume-les-Dames
  - Research Site, Bayonne
  - Research Site, Bâgé-le-Châtel
  - Research Site, Beaucaire
  - Research Site, Beaucouzé
  - Research Site, Beaumont
  - Research Site, Beaumont-de-Pertuis
  - Research Site, Beaumont-lès-Valence
  - Research Site, Beaune
  - Research Site, Beauregard-l'Évêque
  - Research Site, Beausoleil
  - Research Site, Beauvais
  - Research Site, Beauzelle
  - Research Site, Belfort
  - Research Site, Belgodère
  - Research Site, Bellac
  - Research Site, Belleneuve
  - Research Site, Belleville-sur-Meuse
  - Research Site, Bellême
  - Research Site, Belz
  - Research Site, Benfeld
  - Research Site, Bergerac
  - Research Site, Bergholtz
  - Research Site, Berre-l'Étang
  - Research Site, Bersée
  - Research Site, Berson
  - Research Site, Besançon
  - Research Site, Bessé-sur-Braye
  - Research Site, Bessines SUR Gartemp
  - Research Site, Beuvillers
  - Research Site, Beuvry
  - Research Site, Bécon-les-Granits
  - Research Site, Bégard
  - Research Site, Bérat
  - Research Site, Béville-le-Comte
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Billom
  - Research Site, Billy-Montigny
  - Research Site, Billy-sur-Aisne
  - Research Site, Bischheim
  - Research Site, Bizanos
  - Research Site, Bize-Minervois
  - Research Site, Blaesheim
  - Research Site, Blanquefort
  - Research Site, Blaye
  - Research Site, Blenod LES PONT A MO
  - Research Site, Blérancourt
  - Research Site, Blois
  - Research Site, Blotzheim
  - Research Site, Bobigny
  - Research Site, Boeil-Bezing
  - Research Site, Boën-sur-Lignon
  - Research Site, Bois-Colombes
  - Research Site, Bois-Guillaume
  - Research Site, Bois-le-Roi
  - Research Site, Boiscommun
  - Research Site, Boisseuil
  - Research Site, Bolbec
  - Research Site, Bompas
  - Research Site, Bon-Encontre
  - Research Site, Bondy
  - Research Site, Bonneval
  - Research Site, Boos
  - Research Site, Bordeaux
  - Research Site, Bordères-sur-l'Échez
  - Research Site, Bormes-les-Mimosas
  - Research Site, Bort-les-Orgues
  - Research Site, Boucau
  - Research Site, Bouffémont
  - Research Site, Bouguenais
  - Research Site, Boujan-sur-Libron
  - Research Site, Boulbon
  - Research Site, Boulogne-Billancourt
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourg-Achard
  - Research Site, Bourg-de-Péage
  - Research Site, Bourg-des-Comptes
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourg-la-Reine
  - Research Site, Bourg-Lastic
  - Research Site, Bourg-lès-Valence
  - Research Site, Bourges
  - Research Site, Bourron-Marlotte
  - Research Site, Boussac
  - Research Site, Boussy-Saint-Antoine
  - Research Site, Brancourt-le-Grand
  - Research Site, Branne
  - Research Site, Brax
  - Research Site, Bray-sur-Seine
  - Research Site, Brest
  - Research Site, Breteuil
  - Research Site, Brezolles
  - Research Site, Brégnier-Cordon
  - Research Site, Brie
  - Research Site, Brie-Comte-Robert
  - Research Site, Brillac
  - Research Site, Brimeux
  - Research Site, Brion-près-Thouet
  - Research Site, Briouze
  - Research Site, Brives-Charensac
  - Research Site, Bron
  - Research Site, Brou
  - Research Site, Brouvelieures
  - Research Site, Broût-Vernet
  - Research Site, Bruay-la-Buissière
  - Research Site, Bruay-sur-l'Escaut
  - Research Site, Bruges
  - Research Site, Buc
  - Research Site, Buchelay
  - Research Site, Buchy
  - Research Site, Bucy-le-Long
  - Research Site, Bulgnéville
  - Research Site, Bures-sur-Yvette
  - Research Site, Cabannes
  - Research Site, Cachan
  - Research Site, Cadaujac
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cahors
  - Research Site, Calais
  - Research Site, Callac de Bretagne
  - Research Site, Caluire-et-Cuire
  - Research Site, Cambes
  - Research Site, Cambrai
  - Research Site, Cambremer
  - Research Site, Camon
  - Research Site, Campan
  - Research Site, Campbon
  - Research Site, Camphin EN Carembaul
  - Research Site, Canet-en-Roussillon
  - Research Site, Cannes
  - Research Site, Cannes-Écluse
  - Research Site, Canteleu
  - Research Site, Capbreton
  - Research Site, Capdenac-Gare
  - Research Site, Capestang
  - Research Site, Cappelle-en-Pévèle
  - Research Site, Cappelle-la-Grande
  - Research Site, Carantec
  - Research Site, Carcassonne
  - Research Site, Carentan
  - Research Site, Carignan
  - Research Site, Carnac
  - Research Site, Carnoux-en-Provence
  - Research Site, Caromb
  - Research Site, Carpentras
  - Research Site, Carquefou
  - Research Site, Carresse-Cassaber
  - Research Site, Cartignies
  - Research Site, Carvin
  - Research Site, Cassel
  - Research Site, Cassis
  - Research Site, Castanet Tolosan CED
  - Research Site, Castelnau-de-Guers
  - Research Site, Castelnau-le-Lez
  - Research Site, Castelnau-Montratier
  - Research Site, Castres
  - Research Site, Caulnes
  - Research Site, Cauterets
  - Research Site, Cavaillon
  - Research Site, Caylus
  - Research Site, Cendras
  - Research Site, Cenon
  - Research Site, Cergy
  - Research Site, Cergy-Pontoise
  - Research Site, Cervione
  - Research Site, Cesson-Sévigné
  - Research Site, Cérans-Foulletourte
  - Research Site, Cérences
  - Research Site, Cérilly
  - Research Site, Chabris
  - Research Site, Chalabre
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Chambon-sur-Voueize
  - Research Site, Chamonix
  - Research Site, Champagne AU MONT D
  - Research Site, Champagne-sur-Oise
  - Research Site, Champagné-les-Marais
  - Research Site, Champcueil
  - Research Site, Champigny-sur-Marne
  - Research Site, Champniers
  - Research Site, Champs-sur-Marne
  - Research Site, Chanac
  - Research Site, Chanceaux SUR Choisi
  - Research Site, Chanteheux
  - Research Site, Chantepie
  - Research Site, Chantonnay
  - Research Site, Chaource
  - Research Site, Chaptelat
  - Research Site, Charenton-le-Pont
  - Research Site, Charleville-Mézières
  - Research Site, Charmes
  - Research Site, Chasselay
  - Research Site, Chasseneuil DU Poito
  - Research Site, Chateauneuf SUR CHAR
  - Research Site, Chatou
  - Research Site, Chauché
  - Research Site, Chaufour-Notre-Dame
  - Research Site, Chaumes-en-Brie
  - Research Site, Chaumont
  - Research Site, Chauvigny
  - Research Site, Châbons
  - Research Site, Châlons-en-Champagne
  - Research Site, Château-d'Olonne
  - Research Site, Château-la-Vallière
  - Research Site, Château-Thierry
  - Research Site, Châteaubourg
  - Research Site, Châteaudun
  - Research Site, Châteaugay
  - Research Site, Châteaugiron
  - Research Site, Châteaurenard
  - Research Site, Châteauroux
  - Research Site, Châtel-Guyon
  - Research Site, Châtel-Montagne
  - Research Site, Châtelaillon-Plage
  - Research Site, Châtellerault
  - Research Site, Châtelus-Malvaleix
  - Research Site, Châtenay-Malabry
  - Research Site, Châtenois
  - Research Site, Châtenois-les-Forges
  - Research Site, Châtillon
  - Research Site, Châtillon-sur-Seine
  - Research Site, Chennevieres SUR MAR
  - Research Site, Chenôve
  - Research Site, Cherbourg Octeville
  - Research Site, Cheval-Blanc
  - Research Site, Chevannes
  - Research Site, Chevigny-Saint-Sauveur
  - Research Site, Chécy
  - Research Site, Chilleurs-aux-Bois
  - Research Site, Chinon
  - Research Site, Choisey
  - Research Site, Choisy-en-Brie
  - Research Site, Cholet
  - Research Site, Ciboure
  - Research Site, Clairac
  - Research Site, Claix
  - Research Site, Claye-Souilly
  - Research Site, Clermont
  - Research Site, Clermont-Ferrand
  - Research Site, Clérieux
  - Research Site, Clichy
  - Research Site, Clichy-sous-Bois
  - Research Site, Clouange
  - Research Site, Cognac
  - Research Site, Colleville Montgomer
  - Research Site, Collioure
  - Research Site, Colmar
  - Research Site, Colombes
  - Research Site, Colomiers
  - Research Site, Combles
  - Research Site, Combrit
  - Research Site, Combs-la-Ville
  - Research Site, Concarneau
  - Research Site, Conflans STE Honorin
  - Research Site, Conflans-en-Jarnisy
  - Research Site, Conty
  - Research Site, Corbehem
  - Research Site, Corbeil-Essonnes
  - Research Site, Corcieux
  - Research Site, Corme-Royal
  - Research Site, Cormeilles EN Parisi
  - Research Site, Cormicy
  - Research Site, Cornil
  - Research Site, Coubron
  - Research Site, Couches
  - Research Site, Coudekerque-Branche
  - Research Site, Coudes
  - Research Site, Coudun
  - Research Site, Coufouleux
  - Research Site, Coulommiers
  - Research Site, Courbevoie
  - Research Site, Courcelles-sur-Nied
  - Research Site, Courçon
  - Research Site, Cournon-d'Auvergne
  - Research Site, Cours-de-Pile
  - Research Site, Courseulles-sur-Mer
  - Research Site, Courtenay
  - Research Site, Coussac-Bonneval
  - Research Site, Coutances
  - Research Site, Couzon-au-Mont-d'Or
  - Research Site, Cransac
  - Research Site, Craon
  - Research Site, Creil
  - Research Site, Creully
  - Research Site, Creutzwald
  - Research Site, Crèvecœur-le-Grand
  - Research Site, Crécy-sur-Serre
  - Research Site, Crégy-lès-Meaux
  - Research Site, Créhange
  - Research Site, Crépy-en-Valois
  - Research Site, Créteil
  - Research Site, Croissy-sur-Seine
  - Research Site, Croix
  - Research Site, Crolles
  - Research Site, Cros-de-Cagnes
  - Research Site, Crosne
  - Research Site, Cubzac-les-Ponts
  - Research Site, Cugand
  - Research Site, Cugnaux
  - Research Site, Cuincy
  - Research Site, Culoz
  - Research Site, Cusset
  - Research Site, Dainville
  - Research Site, Damas-et-Bettegney
  - Research Site, Dambach-la-Ville
  - Research Site, Dammartin-en-Goële
  - Research Site, Dangé-Saint-Romain
  - Research Site, Darnétal
  - Research Site, Davézieux
  - Research Site, Delle
  - Research Site, Deuil-la-Barre
  - Research Site, Décines-Charpieu
  - Research Site, Déville-lès-Rouen
  - Research Site, Diebling
  - Research Site, Digne-les-Bains
  - Research Site, Dijon
  - Research Site, Dole
  - Research Site, Domène
  - Research Site, Domont
  - Research Site, Dompierre-les-Ormes
  - Research Site, Dompierre-sur-Helpe
  - Research Site, Donges
  - Research Site, Dordives
  - Research Site, Dormans
  - Research Site, Douai
  - Research Site, Douarnenez
  - Research Site, Doubs
  - Research Site, Douchy-les-Mines
  - Research Site, Douelle
  - Research Site, Doué-la-Fontaine
  - Research Site, Dourdan
  - Research Site, Douvres LA Delivrand
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Draveil
  - Research Site, Droué
  - Research Site, Duclair
  - Research Site, Dun-le-Palestel
  - Research Site, Dunkirk
  - Research Site, Duppigheim
  - Research Site, Durtal
  - Research Site, Eaubonne
  - Research Site, Eaunes
  - Research Site, Eauze
  - Research Site, Eckwersheim
  - Research Site, Enghien-les-Bains
  - Research Site, Entrammes
  - Research Site, Envermeu
  - Research Site, Ermont
  - Research Site, Ernée
  - Research Site, Esbly
  - Research Site, Eslettes
  - Research Site, Esquerdes
  - Research Site, Estivareilles
  - Research Site, Eyguières
  - Research Site, Eyragues
  - Research Site, Eyrans
  - Research Site, Eysines
  - Research Site, Èze
  - Research Site, Échirolles
  - Research Site, Éguzon-Chantôme
  - Research Site, Élancourt
  - Research Site, Épernay
  - Research Site, Épernon
  - Research Site, Épinal
  - Research Site, Épinay-sur-Orge
  - Research Site, Épinay-sur-Seine
  - Research Site, Épron
  - Research Site, Étain
  - Research Site, Étretat
  - Research Site, Évin-Malmaison
  - Research Site, Évreux
  - Research Site, Évry-Grégy-sur-Yerre
  - Research Site, Faches-Thumesnil
  - Research Site, Fameck
  - Research Site, Fampoux
  - Research Site, Faverges
  - Research Site, Feignies
  - Research Site, Fenouillet
  - Research Site, Fesches-le-Châtel
  - Research Site, Feuchy
  - Research Site, Feurs
  - Research Site, Feyzin
  - Research Site, Fécamp
  - Research Site, Figeac
  - Research Site, Fillinges
  - Research Site, Finhan
  - Research Site, Firminy
  - Research Site, Flavin
  - Research Site, Flers
  - Research Site, Flers-en-Escrebieux
  - Research Site, Flesselles
  - Research Site, Fleury-les-Aubrais
  - Research Site, Fleville Devant NANC
  - Research Site, Flize
  - Research Site, Folembray
  - Research Site, Fonbeauzard
  - Research Site, Fontaine
  - Research Site, Fontaine-le-Comte
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Fontainebleau
  - Research Site, Fontanil-Cornillon
  - Research Site, Fontenay-sous-Bois
  - Research Site, Forbach
  - Research Site, Fos-sur-Mer
  - Research Site, Fougères
  - Research Site, Fouras
  - Research Site, Fourneaux
  - Research Site, Francescas
  - Research Site, Franconville LA GARE
  - Research Site, Frasne
  - Research Site, Fresnes-en-Woëvre
  - Research Site, Fréjus
  - Research Site, Fronsac
  - Research Site, Frouard
  - Research Site, Furiani
  - Research Site, Gagny
  - Research Site, Gaillon
  - Research Site, Gainneville
  - Research Site, Gallardon
  - Research Site, Gambsheim
  - Research Site, Gannat
  - Research Site, Gap
  - Research Site, Gardanne
  - Research Site, Gargenville
  - Research Site, Garges-lès-Gonesse
  - Research Site, Gasny
  - Research Site, Gauchy
  - Research Site, Gazinet
  - Research Site, Gelos
  - Research Site, Gençay
  - Research Site, Geneuille
  - Research Site, Genillé
  - Research Site, Gennevilliers
  - Research Site, Gentilly
  - Research Site, Gerbéviller
  - Research Site, Gex
  - Research Site, Gien
  - Research Site, Gif-sur-Yvette
  - Research Site, Gignac
  - Research Site, Girmont
  - Research Site, Goncelin
  - Research Site, Gondrecourt LE Chate
  - Research Site, Gondreville
  - Research Site, Gorcy
  - Research Site, Gorron
  - Research Site, Gourdon
  - Research Site, Gouzon
  - Research Site, Gramat
  - Research Site, Grambois
  - Research Site, Granville
  - Research Site, Grasse
  - Research Site, Graulhet
  - Research Site, Grenade
  - Research Site, Grenoble
  - Research Site, Gréasque
  - Research Site, Grésy-sur-Aix
  - Research Site, Grésy-sur-Isère
  - Research Site, Grièges
  - Research Site, Guarbecque
  - Research Site, Guebwiller
  - Research Site, Guessling-Hémering
  - Research Site, Guénange
  - Research Site, Guéreins
  - Research Site, Guéret
  - Research Site, Guidel
  - Research Site, Guipavas
  - Research Site, Guipel
  - Research Site, Guipry
  - Research Site, Guise
  - Research Site, Guitalens-L'Albarède
  - Research Site, Guyancourt
  - Research Site, Gy
  - Research Site, Haguenau
  - Research Site, Haillicourt
  - Research Site, Hallennes LEZ Haubou
  - Research Site, Halluin
  - Research Site, Hanvec
  - Research Site, Hardelot-Plage
  - Research Site, Haspres
  - Research Site, Haut-Mauco
  - Research Site, Hautmont
  - Research Site, Hazebrouck
  - Research Site, Hellemmes-Lille
  - Research Site, Hendaye
  - Research Site, Hennebont
  - Research Site, Herbault
  - Research Site, Hénin-Beaumont
  - Research Site, Héricourt-en-Caux
  - Research Site, Hérouville-Saint-Clair
  - Research Site, Holnon
  - Research Site, Honfleur
  - Research Site, Horbourg-Wihr
  - Research Site, Houilles
  - Research Site, Houplin-Ancoisne
  - Research Site, Hourtin
  - Research Site, Hulluch
  - Research Site, Hurigny
  - Research Site, Hyères
  - Research Site, Hœrdt
  - Research Site, Igé
  - Research Site, Illkirch Graffenstad
  - Research Site, Inchy
  - Research Site, Ingrandes
  - Research Site, Is-sur-Tille
  - Research Site, Isbergues
  - Research Site, Issy-les-Moulineaux
  - Research Site, Istres
  - Research Site, Ivoy-le-Pré
  - Research Site, Ivry-sur-Seine
  - Research Site, Jassans-Riottier
  - Research Site, Jaunay-Clan
  - Research Site, Jeumont
  - Research Site, Joinville-le-Pont
  - Research Site, Jonchery-sur-Vesle
  - Research Site, Jonquières
  - Research Site, Jouars-Pontchartrain
  - Research Site, Joué-lès-Tours
  - Research Site, Joze
  - Research Site, Juan-les-Pins
  - Research Site, Jurançon
  - Research Site, Jussey
  - Research Site, Juvignac
  - Research Site, Juvigné
  - Research Site, Kerbach
  - Research Site, Kersaint-Plabennec
  - Research Site, Kurtzenhouse
  - Research Site, L'Aigle
  - Research Site, L'Étrat
  - Research Site, L'Horme
  - Research Site, L'Huisserie
  - Research Site, L'Isle-d'Abeau
  - Research Site, L'Isle-en-Dodon
  - Research Site, L'Isle-Jourdain
  - Research Site, L'Isle-sur-la-Sorgue
  - Research Site, L'Île-d'Olonne
  - Research Site, L'Île-Rousse
  - Research Site, L'Île-Saint-Denis
  - Research Site, La Balme-de-Sillingy
  - Research Site, La Bassée
  - Research Site, La Bouëxière
  - Research Site, La Bouilladisse
  - Research Site, La Celle-Saint-Cloud
  - Research Site, La Chapelaude
  - Research Site, LA Chapelle DES FOUG
  - Research Site, LA Chapelle DES MARA
  - Research Site, LA Chaussee SUR MARN
  - Research Site, La Ciotat
  - Research Site, La Colle-sur-Loup
  - Research Site, La Coquille
  - Research Site, La Courneuve
  - Research Site, La Couronne
  - Research Site, La Crau
  - Research Site, LA Ferriere AUX ETAN
  - Research Site, La Ferrière
  - Research Site, La Ferté-Imbault
  - Research Site, La Ferté-Macé
  - Research Site, La Ferté-Saint-Aubin
  - Research Site, La Fouillade
  - Research Site, La Garde
  - Research Site, La Garenne-Colombes
  - Research Site, La Garnache
  - Research Site, La Gaude
  - Research Site, La Grand-Combe
  - Research Site, La Grand-Croix
  - Research Site, LA Guerche SUR L AUB
  - Research Site, La Jaudonnière
  - Research Site, La Jubaudière
  - Research Site, La Londe-les-Maures
  - Research Site, La Loupe
  - Research Site, La Madeleine
  - Research Site, LA Mailleraye SUR SE
  - Research Site, La Motte-Servolex
  - Research Site, La Mulatière
  - Research Site, La Mure
  - Research Site, La Queue-en-Brie
  - Research Site, La Réole
  - Research Site, La Roche-en-Brenil
  - Research Site, La Roche-Posay
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochefoucauld
  - Research Site, La Rochelle
  - Research Site, LA Seyne SUR MER CED
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Talaudière
  - Research Site, La Tour-de-Salvagny
  - Research Site, La Turballe
  - Research Site, La Turbie
  - Research Site, LA Varenne Saint Hilair
  - Research Site, La Verpillière
  - Research Site, Labastide-Murat
  - Research Site, Labastide-Saint-Georges
  - Research Site, Labastidette
  - Research Site, Labruguière
  - Research Site, Lafox
  - Research Site, Lagarde-Enval
  - Research Site, Lagardelle-sur-Lèze
  - Research Site, Lagnieu
  - Research Site, Lagny-sur-Marne
  - Research Site, Lagord
  - Research Site, Laissac
  - Research Site, Lamagistère
  - Research Site, Lamballe
  - Research Site, Lambersart
  - Research Site, Lamonzie
  - Research Site, Lamorlaye
  - Research Site, Lampertheim
  - Research Site, Landerneau
  - Research Site, Landivisiau
  - Research Site, Landivy
  - Research Site, Langeac
  - Research Site, Langeais
  - Research Site, Langonnet
  - Research Site, Lanildut
  - Research Site, Lanmeur
  - Research Site, Lannemezan
  - Research Site, Lanouée
  - Research Site, Lanton
  - Research Site, Laragne-Montéglin
  - Research Site, LArbresle
  - Research Site, Larmor-Plage
  - Research Site, Lassigny
  - Research Site, Lathus-Saint-Rémy
  - Research Site, Latresne
  - Research Site, Lattes
  - Research Site, Laudun-lArdoise
  - Research Site, Laure
  - Research Site, Lauterbourg
  - Research Site, Laval
  - Research Site, Lavardac
  - Research Site, Lavaveix-les-Mines
  - Research Site, Lavernose-Lacasse
  - Research Site, Lavit
  - Research Site, Laxou
  - Research Site, Le Ban Saint-Martin
  - Research Site, Le Blanc-Mesnil
  - Research Site, Le Bourget
  - Research Site, Le Bourget-du-Lac
  - Research Site, Le Bouscat
  - Research Site, Le Cannet
  - Research Site, Le Cap D'Agde
  - Research Site, Le Cendre
  - Research Site, Le Chesnay
  - Research Site, Le Coudray-Montceaux
  - Research Site, Le Crès
  - Research Site, Le Croisic
  - Research Site, Le Fleix
  - Research Site, Le Folgoët
  - Research Site, Le Gâvre
  - Research Site, LE Golfe JUAN
  - Research Site, Le Grand-Lucé
  - Research Site, Le Grand-Quevilly
  - Research Site, Le Havre
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Lion-dAngers
  - Research Site, Le Louroux Béconnais
  - Research Site, Le Mans
  - Research Site, Le Mas-d'Agenais
  - Research Site, Le May-sur-Èvre
  - Research Site, Le Mesnil-Esnard
  - Research Site, Le Mée-sur-Seine
  - Research Site, Le Mêle-sur-Sarthe
  - Research Site, LE Monastier SUR GAZ
  - Research Site, Le Passage
  - Research Site, LE Perray EN Yveline
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Petit-Quevilly
  - Research Site, Le Plan-de-Grasse
  - Research Site, Le Plessis-Trévise
  - Research Site, Le Poiré-sur-Vie
  - Research Site, Le Pontet
  - Research Site, Le Port-Marly
  - Research Site, Le Pouliguen
  - Research Site, Le Pradet
  - Research Site, Le Relecq-Kerhuon
  - Research Site, Le Revest-les-Eaux
  - Research Site, Le Rheu
  - Research Site, Le Russey
  - Research Site, Le Soler
  - Research Site, Le Teil
  - Research Site, LE Touquet Paris PLA
  - Research Site, Le Verdon-sur-Mer
  - Research Site, Le Vésinet
  - Research Site, Le Vigen
  - Research Site, Lectoure
  - Research Site, Lempdes
  - Research Site, Lens
  - Research Site, Les Andelys
  - Research Site, Les Clayes-sous-Bois
  - Research Site, LES Contamines Montj
  - Research Site, Les Essarts
  - Research Site, LES Eyzies Tayac SIR
  - Research Site, Les Échelles
  - Research Site, Les Issambres
  - Research Site, Les Lilas
  - Research Site, Les Montils
  - Research Site, Les Mureaux
  - Research Site, Les Ormes
  - Research Site, LES Pavillons SOUS B
  - Research Site, Lesconil
  - Research Site, Levallois-Perret
  - Research Site, Lécluse
  - Research Site, Lédignan
  - Research Site, Lérouville
  - Research Site, Léry
  - Research Site, Lévignac
  - Research Site, Lézardrieux
  - Research Site, Lézignan-Corbières
  - Research Site, LIEU DIT Carnon PLAG
  - Research Site, Liévin
  - Research Site, Liffol-le-Grand
  - Research Site, Liffré
  - Research Site, Ligny-en-Cambrésis
  - Research Site, Lille
  - Research Site, Lillebonne
  - Research Site, Limas
  - Research Site, Limay
  - Research Site, Limeray
  - Research Site, Limoges
  - Research Site, Limogne-en-Quercy
  - Research Site, Linas
  - Research Site, Lingolsheim
  - Research Site, Lisses
  - Research Site, Livron-sur-Drôme
  - Research Site, Livry-Gargan
  - Research Site, Lizy-sur-Ourcq
  - Research Site, Loison-sous-Lens
  - Research Site, Lombez
  - Research Site, Lomme
  - Research Site, Longueau
  - Research Site, Longueville
  - Research Site, Longué-Jumelles
  - Research Site, Lons-le-Saunier
  - Research Site, Loon-Plage
  - Research Site, Loos
  - Research Site, Loos-en-Gohelle
  - Research Site, Loperhet
  - Research Site, Lorgues
  - Research Site, Lormont
  - Research Site, Lourdes
  - Research Site, Louveciennes
  - Research Site, Louviers
  - Research Site, Louvigné-de-Bais
  - Research Site, Louvigné-du-Désert
  - Research Site, Lucé
  - Research Site, Luçon
  - Research Site, Lumes
  - Research Site, Lunéville
  - Research Site, Lurcy-Lévis
  - Research Site, Lury-sur-Arnon
  - Research Site, Lusigny
  - Research Site, Lussac-les-Églises
  - Research Site, Luxeuil-les-Bains
  - Research Site, Lyon
  - Research Site, L’Isle-sur-le-Doubs
  - Research Site, Mably
  - Research Site, Madonne-et-Lamerey
  - Research Site, Maël-Carhaix
  - Research Site, Magalas
  - Research Site, Magland
  - Research Site, Magny-les-Hameaux
  - Research Site, Maillot
  - Research Site, Mailly-Maillet
  - Research Site, Maintenon
  - Research Site, Maisons-Alfort
  - Research Site, Maisons-Laffitte
  - Research Site, Malemort-du-Comtat
  - Research Site, Malemort-sur-Corrèze
  - Research Site, Malesherbes
  - Research Site, Malestroit
  - Research Site, Malo-les-Bains
  - Research Site, Mamers
  - Research Site, Manciet
  - Research Site, Mancieulles
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Manosque
  - Research Site, Mantes-la-Jolie
  - Research Site, Marange-Silvange
  - Research Site, Marchiennes
  - Research Site, Marcilly-en-Villette
  - Research Site, Mareuil SUR LAY DISS
  - Research Site, Marguerittes
  - Research Site, Marignane
  - Research Site, Marigny-le-Châtel
  - Research Site, Maringues
  - Research Site, Marles-les-Mines
  - Research Site, Marly
  - Research Site, Marmande
  - Research Site, Maromme
  - Research Site, Marquion
  - Research Site, Marsannay-la-Côte
  - Research Site, Marsas
  - Research Site, Marseille
  - Research Site, Marspich
  - Research Site, Martigues
  - Research Site, Martin-Église
  - Research Site, Marvejols
  - Research Site, Matha
  - Research Site, Mathay
  - Research Site, Mathieu
  - Research Site, Maubeuge
  - Research Site, Mauguio
  - Research Site, Maule
  - Research Site, Maurepas
  - Research Site, Mauriac
  - Research Site, Maurs
  - Research Site, Mauvezin
  - Research Site, Mauzé-sur-le-Mignon
  - Research Site, Mayenne
  - Research Site, Meaux
  - Research Site, Meillonnas
  - Research Site, Mellecey
  - Research Site, Mennecy
  - Research Site, Mens
  - Research Site, Menton
  - Research Site, Mer
  - Research Site, Mers-les-Bains
  - Research Site, Merville
  - Research Site, Messei
  - Research Site, Messery
  - Research Site, Metz
  - Research Site, Meudon
  - Research Site, Meulan-en-Yvelines
  - Research Site, Meusnes
  - Research Site, Meximieux
  - Research Site, Meylan
  - Research Site, Meyzieu
  - Research Site, Médis
  - Research Site, Médréac
  - Research Site, Méréville
  - Research Site, Mérignac
  - Research Site, Mérindol
  - Research Site, Mézidon-Canon
  - Research Site, Migennes
  - Research Site, Milhaud
  - Research Site, Millas
  - Research Site, Mimet
  - Research Site, Mions
  - Research Site, Mirabeau
  - Research Site, Miramont-de-Guyenne
  - Research Site, Mirecourt
  - Research Site, Miribel-les-Échelles
  - Research Site, Mitry-Mory
  - Research Site, Moëlan-sur-Mer
  - Research Site, Moissac
  - Research Site, Molsheim
  - Research Site, Moncé-en-Belin
  - Research Site, Mondeville
  - Research Site, Mondragon
  - Research Site, Monéteau
  - Research Site, Mons-en-Barœul
  - Research Site, Monswiller
  - Research Site, Mont-Saint-Aignan
  - Research Site, Montady
  - Research Site, Montaren ET Saint Medie
  - Research Site, Montauban
  - Research Site, Montbazin
  - Research Site, Montbéliard
  - Research Site, Montbonnot-Saint-Martin
  - Research Site, Montbrison
  - Research Site, Montceau-les-Mines
  - Research Site, Montcy-Notre-Dame
  - Research Site, Montendre
  - Research Site, Montesson
  - Research Site, Montfermeil
  - Research Site, Montferrat
  - Research Site, Montfrin
  - Research Site, Montgeron
  - Research Site, Montigny-lès-Metz
  - Research Site, Montigny-sur-Loing
  - Research Site, Montivilliers
  - Research Site, Montlieu-la-Garde
  - Research Site, Montluçon
  - Research Site, Montluel
  - Research Site, Montmagny
  - Research Site, Montmorillon
  - Research Site, Montoir-de-Bretagne
  - Research Site, Montoison
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montreuil-l'Argillé
  - Research Site, Montrevel-en-Bresse
  - Research Site, Montrouge
  - Research Site, Morcenx
  - Research Site, Mordelles
  - Research Site, Moret-sur-Loing
  - Research Site, Moreuil
  - Research Site, Morhange
  - Research Site, Morlaàs
  - Research Site, Mornant
  - Research Site, Morre
  - Research Site, Morsang-sur-Orge
  - Research Site, Mortagne-sur-Gironde
  - Research Site, Mortain
  - Research Site, Morteau
  - Research Site, Mouchin
  - Research Site, Moulins-lès-Metz
  - Research Site, Mourmelon-le-Petit
  - Research Site, Moutiers LES Mauxfai
  - Research Site, Mouvaux
  - Research Site, Mouy
  - Research Site, Moyeuvre-Grande
  - Research Site, Mulhouse
  - Research Site, Muret
  - Research Site, Mussidan
  - Research Site, Nailhac
  - Research Site, Naintré
  - Research Site, Nalliers
  - Research Site, Nancy
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Nasbinals
  - Research Site, Naucelles
  - Research Site, Naveil
  - Research Site, Nay
  - Research Site, Neauphle-le-Château
  - Research Site, Nemours
  - Research Site, Neuillé-Pont-Pierre
  - Research Site, Neuilly-lès-Dijon
  - Research Site, Neuilly-sur-Marne
  - Research Site, Neuilly-sur-Seine
  - Research Site, Neulise
  - Research Site, Neuves-Maisons
  - Research Site, Neuville-de-Poitou
  - Research Site, Neuville-en-Ferrain
  - Research Site, Neuville-lès-Dieppe
  - Research Site, Neuvy-Pailloux
  - Research Site, Nevers
  - Research Site, Nexon
  - Research Site, Nègrepelisse
  - Research Site, Nice
  - Research Site, Niederschaeffolsheim
  - Research Site, Nieul
  - Research Site, Nilvange
  - Research Site, Nîmes
  - Research Site, Nogent-le-Rotrou
  - Research Site, Nogent-sur-Oise
  - Research Site, Noisy-le-Grand
  - Research Site, Nomeny
  - Research Site, Notre-Dame-de-Riez
  - Research Site, Nouâtre
  - Research Site, Noves
  - Research Site, Noyelles-Godault
  - Research Site, Noyelles-sous-Lens
  - Research Site, Noyers-sur-Cher
  - Research Site, Nuisement-sur-Coole
  - Research Site, Nœux-les-Mines
  - Research Site, Obernai
  - Research Site, Oignies
  - Research Site, Olby
  - Research Site, Olivet
  - Research Site, Olonzac
  - Research Site, Ondres
  - Research Site, Onnaing
  - Research Site, Oradour-sur-Vayres
  - Research Site, Oraison
  - Research Site, Orchamps-Vennes
  - Research Site, Orgeval
  - Research Site, Orléans
  - Research Site, Ormoy
  - Research Site, Orry-la-Ville
  - Research Site, Orthez
  - Research Site, Orvault
  - Research Site, Ostwald
  - Research Site, Oudon
  - Research Site, Ouistreham
  - Research Site, Ouroux-sur-Saône
  - Research Site, Pacé
  - Research Site, Pagny-sur-Moselle
  - Research Site, Pamiers
  - Research Site, Pantin
  - Research Site, Parcé-sur-Sarthe
  - Research Site, Pardies
  - Research Site, Paris
  - Research Site, Parthenay
  - Research Site, Pau
  - Research Site, Peltre
  - Research Site, Percy
  - Research Site, Perpignan
  - Research Site, Perrigny
  - Research Site, Perros-Guirec
  - Research Site, Perrusson
  - Research Site, Persac
  - Research Site, Perthes
  - Research Site, Pertuis
  - Research Site, Pessac
  - Research Site, Petit-Couronne
  - Research Site, Peynier
  - Research Site, Pénestin
  - Research Site, Périgueux
  - Research Site, Péronnas
  - Research Site, Péronne
  - Research Site, Pfaffenhoffen
  - Research Site, Pfetterhouse
  - Research Site, Pierrefitte SUR SAUL
  - Research Site, Pierrefitte SUR SEIN
  - Research Site, Pierrelaye
  - Research Site, Pierrepont-sur-Avre
  - Research Site, Pipriac
  - Research Site, Plaimpied-Givaudins
  - Research Site, Plaisir
  - Research Site, Plan-de-Cuques
  - Research Site, Plascassier
  - Research Site, Pleaux
  - Research Site, Plessala
  - Research Site, Pleubian
  - Research Site, Pleumeur-Bodou
  - Research Site, Pléhédel
  - Research Site, Ploemeur
  - Research Site, Ploërmel
  - Research Site, Plouénan
  - Research Site, Ploumagoar
  - Research Site, Plourhan
  - Research Site, Plouvorn
  - Research Site, Plouzané
  - Research Site, Pluvigner
  - Research Site, Poissy
  - Research Site, Poitiers
  - Research Site, Poligny
  - Research Site, PONT STE Maxence
  - Research Site, Pont-Audemer
  - Research Site, Pont-Aven
  - Research Site, Pont-à-Marcq
  - Research Site, Pont-à-Mousson
  - Research Site, Pont-de-l'Arche
  - Research Site, Pont-de-Roide
  - Research Site, Pont-de-Salars
  - Research Site, Pont-Évêque
  - Research Site, Pont-Scorff
  - Research Site, Pontarlier
  - Research Site, Pontault-Combault
  - Research Site, Pontivy
  - Research Site, Pornichet
  - Research Site, Port Leucate
  - Research Site, PORT Saint Louis DU RHO
  - Research Site, Port-de-Bouc
  - Research Site, Portes-lès-Valence
  - Research Site, Porto-Vecchio
  - Research Site, Pouilly SOUS Charlie
  - Research Site, Poulx
  - Research Site, Pradines
  - Research Site, Prayssac
  - Research Site, Preignac
  - Research Site, Presles
  - Research Site, Pressac
  - Research Site, Pré-en-Pail
  - Research Site, Préchac
  - Research Site, Prix-lès-Mézières
  - Research Site, Provins
  - Research Site, Puget-sur-Argens
  - Research Site, Puichéric
  - Research Site, Pulnoy
  - Research Site, Pusey
  - Research Site, Puteaux
  - Research Site, Puy-Guillaume
  - Research Site, Quesnoy-sur-Deûle
  - Research Site, Quevauvillers
  - Research Site, Quiberon
  - Research Site, Quiers-sur-Bézonde
  - Research Site, Quiévy
  - Research Site, Quimper
  - Research Site, Quimperlé
  - Research Site, Quincy-sous-Sénart
  - Research Site, Quincy-Voisins
  - Research Site, Quinçay
  - Research Site, Quint-Fonsegrives
  - Research Site, Raismes
  - Research Site, Ramonville-Saint-Agne
  - Research Site, Rauzan
  - Research Site, Rebreuve-Ranchicourt
  - Research Site, Recologne
  - Research Site, Reims
  - Research Site, Remiremont
  - Research Site, Rennes
  - Research Site, Revin
  - Research Site, Rezé
  - Research Site, Ria-Sirach
  - Research Site, Ribecourt Dreslincou
  - Research Site, Ribérac
  - Research Site, Richardménil
  - Research Site, Richebourg
  - Research Site, Riedisheim
  - Research Site, Rieupeyroux
  - Research Site, Rilhac-Rancon
  - Research Site, Riquewihr
  - Research Site, Rive-de-Gier
  - Research Site, Rivehaute
  - Research Site, Rivery
  - Research Site, Robert-Espagne
  - Research Site, Rochefort
  - Research Site, Rodez
  - Research Site, Rodilhan
  - Research Site, Rognac
  - Research Site, Rohrbach-lès-Bitche
  - Research Site, Rohrwiller
  - Research Site, Romagné
  - Research Site, Romainville
  - Research Site, Rombas
  - Research Site, Romillé
  - Research Site, Romilly-sur-Seine
  - Research Site, Romorantin-Lanthenay
  - Research Site, Roncey
  - Research Site, Ronchin
  - Research Site, Roncq
  - Research Site, Roppe
  - Research Site, Roquefort-la-Bédoule
  - Research Site, Rosiers-d'Égletons
  - Research Site, Rosny-sous-Bois
  - Research Site, Rospez
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rouhling
  - Research Site, Roulans
  - Research Site, Rousset
  - Research Site, Royan
  - Research Site, Roye
  - Research Site, Ruaudin
  - Research Site, Rueil-Malmaison
  - Research Site, Ruoms
  - Research Site, Ruy
  - Research Site, Ruynes-en-Margeride
  - Research Site, Saffré
  - Research Site, Sahurs
  - Research Site, Sainghin EN Melantoi
  - Research Site, Sains-du-Nord
  - Research Site, Saint Aubin DES Chateau
  - Research Site, Saint Barthelemy de VAL
  - Research Site, Saint Denis LES Olliere
  - Research Site, Saint ERME Outre ET RAM
  - Research Site, Saint Etienne de Baigor
  - Research Site, Saint Etienne de Montlu
  - Research Site, Saint Etienne de Tulmon
  - Research Site, Saint Etienne DU Rouvra
  - Research Site, Saint Firmin EN Valgode
  - Research Site, Saint Georges de Rouell
  - Research Site, Saint Georges DES Grose
  - Research Site, Saint Germain de Marenc
  - Research Site, Saint Germain LES Corbe
  - Research Site, Saint Lambert LA Pother
  - Research Site, Saint Marcel LES Valenc
  - Research Site, Saint Martin D Hardingh
  - Research Site, Saint Martin de Seignan
  - Research Site, Saint Mathieu de Trevie
  - Research Site, Saint Maximin LA STE BA
  - Research Site, Saint PAUL Trois Chatea
  - Research Site, Saint Philbert de Bouai
  - Research Site, Saint Pierre de Chandie
  - Research Site, Saint Pierre de Mannevi
  - Research Site, Saint Pourcain SUR SIOU
  - Research Site, Saint Quentin LA Poteri
  - Research Site, Saint REMY LES Chevreus
  - Research Site, Saint Romain de Jaliona
  - Research Site, Saint Sauveur LE Vicomt
  - Research Site, Saint Sebastien SUR LOI
  - Research Site, Saint Sulpice ET Cameyr
  - Research Site, Saint-Aigulin
  - Research Site, Saint-Amé
  - Research Site, Saint-André-de-la-Roche
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-André-des-Eaux
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Arnoult-en-Yvelines
  - Research Site, Saint-Astier
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Aunès
  - Research Site, Saint-Avold
  - Research Site, Saint-Beauzire
  - Research Site, Saint-Benoît
  - Research Site, Saint-Blaise-la-Roche
  - Research Site, Saint-Bonnet-le-Château
  - Research Site, Saint-Brevin-les-Pins
  - Research Site, Saint-Brévin-l'Océan
  - Research Site, Saint-Brice-sur-Vienne
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Chaffrey
  - Research Site, Saint-Chamond
  - Research Site, Saint-Christol-les-Alès
  - Research Site, Saint-Coulomb
  - Research Site, Saint-Cyr-l'École
  - Research Site, Saint-Cyr-sur-Mer
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-d'Orques
  - Research Site, Saint-Didier-en-Velay
  - Research Site, Saint-Dié
  - Research Site, Saint-Dizier
  - Research Site, Saint-Etienne
  - Research Site, Saint-Égrève
  - Research Site, Saint-Évarzec
  - Research Site, Saint-Fargeau
  - Research Site, Saint-Féliu-d'Avall
  - Research Site, Saint-Félix-de-Lodez
  - Research Site, Saint-Florent-sur-Cher
  - Research Site, Saint-Flour
  - Research Site, Saint-Fons
  - Research Site, Saint-Gaudens
  - Research Site, Saint-Georges-du-Bois
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Saint-Gervais-en-Belin
  - Research Site, Saint-Gilles
  - Research Site, Saint-Girons
  - Research Site, Saint-Gobain
  - Research Site, Saint-Herblain
  - Research Site, Saint-Hilaire-des-Loges
  - Research Site, Saint-Jean-Bonnefonds
  - Research Site, Saint-Jean-de-la-Ruelle
  - Research Site, Saint-Jean-de-Liversay
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-de-Maurienne
  - Research Site, Saint-Jean-Pied-de-Port
  - Research Site, Saint-Jeannet
  - Research Site, Saint-Jory
  - Research Site, Saint-Julien-de-Civry
  - Research Site, Saint-Julien-les-Villas
  - Research Site, Saint-Just-d'Ardèche
  - Research Site, Saint-Just-Saint-Rambert
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Laurent-sur-Gorre
  - Research Site, Saint-Léger-lès-Domart
  - Research Site, Saint-Loubès
  - Research Site, Saint-Louis
  - Research Site, Saint-Loup-sur-Semouse
  - Research Site, Saint-Lupicin
  - Research Site, Saint-Lyphard
  - Research Site, Saint-Lys
  - Research Site, Saint-Macaire-en-Mauges
  - Research Site, Saint-Mamert-du-Gard
  - Research Site, Saint-Mamet-la-Salvetat
  - Research Site, Saint-Mandé
  - Research Site, Saint-Marcel-sur-Aude
  - Research Site, Saint-Marcellin
  - Research Site, Saint-Martin-d'Hères
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Maurice-des-Lions
  - Research Site, Saint-Médard-en-Jalles
  - Research Site, Saint-Michel-Chef-Chef
  - Research Site, Saint-Mihiel
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Nom-la-Bretêche
  - Research Site, Saint-Paul-en-Jarez
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Paul-lès-Romans
  - Research Site, Saint-Philibert
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pierre-des-Fleurs
  - Research Site, Saint-Pol-sur-Ternoise
  - Research Site, Saint-Porchaire
  - Research Site, Saint-Priest
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Pryvé-Saint-Mesmin
  - Research Site, Saint-Quentin
  - Research Site, Saint-Rambert-d'Albon
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Saint-Romain-de-Colbosc
  - Research Site, Saint-Romain-la-Motte
  - Research Site, Saint-Saëns
  - Research Site, Saint-Sauveur
  - Research Site, Saint-Savinien
  - Research Site, Saint-Savournin
  - Research Site, Saint-Sornin-Leulac
  - Research Site, Saint-Sulpice-de-Royan
  - Research Site, Saint-Thuriau
  - Research Site, Saint-Urbain
  - Research Site, Saint-Vrain
  - Research Site, Saint-Yan
  - Research Site, Saint-Yorre
  - Research Site, Saintes
  - Research Site, Salers
  - Research Site, Saleux
  - Research Site, Salies-du-Salat
  - Research Site, Samer
  - Research Site, Sanary-sur-Mer
  - Research Site, Sannois
  - Research Site, Sarcelles
  - Research Site, Sargé-lès-le-Mans
  - Research Site, Sarre-Union
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Sartrouville
  - Research Site, Sassenage
  - Research Site, Saugnac-et-Cambran
  - Research Site, Saulieu
  - Research Site, Saulzoir
  - Research Site, Sausheim
  - Research Site, Sauveterre de Rouerg
  - Research Site, Sauveterre-de-Béarn
  - Research Site, Savines-le-Lac
  - Research Site, Sayat
  - Research Site, Schiltigheim
  - Research Site, Schirrhein
  - Research Site, Segonzac
  - Research Site, Segré
  - Research Site, Seichamps
  - Research Site, Selles-sur-Cher
  - Research Site, Semblançay
  - Research Site, Semécourt
  - Research Site, Senones
  - Research Site, Sens
  - Research Site, Sens-de-Bretagne
  - Research Site, Sermaises
  - Research Site, Sermoise-sur-Loire
  - Research Site, Sers
  - Research Site, Servian
  - Research Site, Sessenheim
  - Research Site, Sevran
  - Research Site, Seyssins
  - Research Site, Seyssuel
  - Research Site, Sète
  - Research Site, Sélestat
  - Research Site, Séméac
  - Research Site, Sénas
  - Research Site, Sérignan
  - Research Site, Sigean
  - Research Site, Six-Fours-les-Plages
  - Research Site, Sixt-sur-Aff
  - Research Site, Soissons
  - Research Site, Soisy SOUS Montmoren
  - Research Site, Solesmes
  - Research Site, Solliès-Pont
  - Research Site, Somain
  - Research Site, Sommières
  - Research Site, Sonchamp
  - Research Site, Sorbiers
  - Research Site, Sorgues
  - Research Site, Sospel
  - Research Site, Sotteville-lès-Rouen
  - Research Site, Souchez
  - Research Site, Soucy
  - Research Site, Souffelweyersheim
  - Research Site, Soufflenheim
  - Research Site, Souillac
  - Research Site, Soullans
  - Research Site, Soultz-Haut-Rhin
  - Research Site, Soyaux
  - Research Site, St-Malo
  - Research Site, St.-Jean
  - Research Site, Stains
  - Research Site, STE Bazeille
  - Research Site, STE Consorce
  - Research Site, STE Feyre
  - Research Site, STE Florine
  - Research Site, STE Fortunade
  - Research Site, STE FOY de Peyrolier
  - Research Site, STE Genevieve DES BO
  - Research Site, STE Hermine
  - Research Site, STE LUCE SUR Loire
  - Research Site, STE Marie SUR Ouche
  - Research Site, Strasbourg
  - Research Site, Stuckange
  - Research Site, Survilliers
  - Research Site, Talence
  - Research Site, Tarascon
  - Research Site, Tarbes
  - Research Site, Targon
  - Research Site, Tassin-la-Demi-Lune
  - Research Site, Taulignan
  - Research Site, Taverny
  - Research Site, Terminiers
  - Research Site, Teyran
  - Research Site, Thénezay
  - Research Site, Thérondels
  - Research Site, Thizy
  - Research Site, Thonon-les-Bains
  - Research Site, Thorigny-sur-Marne
  - Research Site, Thumeries
  - Research Site, Tigy
  - Research Site, Til-Châtel
  - Research Site, Tilly-sur-Seulles
  - Research Site, Tincques
  - Research Site, Torcy
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tourlaville
  - Research Site, Tournefeuille
  - Research Site, Tournon-sur-Rhône
  - Research Site, Tournus
  - Research Site, Tours
  - Research Site, Tracy-le-Mont
  - Research Site, Traînel
  - Research Site, Trans-en-Provence
  - Research Site, Treize-Vents
  - Research Site, Trets
  - Research Site, Trégueux
  - Research Site, Trélazé
  - Research Site, Trévières
  - Research Site, Tricot
  - Research Site, Trieux
  - Research Site, Trignac
  - Research Site, Troarn
  - Research Site, Troo
  - Research Site, Troyes
  - Research Site, Turretot
  - Research Site, Urt
  - Research Site, Uxem
  - Research Site, Vabres-l'Abbaye
  - Research Site, Vailly-sur-Aisne
  - Research Site, Valberg
  - Research Site, Valbonne
  - Research Site, Valdoie
  - Research Site, Valence
  - Research Site, Valensole
  - Research Site, Valenton
  - Research Site, Vallauris
  - Research Site, Vallières
  - Research Site, Vallon-sur-Gée
  - Research Site, Valmondois
  - Research Site, Valmont
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vannes
  - Research Site, Varangéville
  - Research Site, Varennes-Vauzelles
  - Research Site, Vaugneray
  - Research Site, Vaulx-en-Velin
  - Research Site, Veigné
  - Research Site, Velaux
  - Research Site, Velleron
  - Research Site, Venarey-les-Laumes
  - Research Site, Vendôme
  - Research Site, Venerque
  - Research Site, Vennecy
  - Research Site, Ventabren
  - Research Site, Verdun
  - Research Site, Verdun-sur-Garonne
  - Research Site, Vernouillet
  - Research Site, Verny
  - Research Site, Vers-Pont-du-Gard
  - Research Site, Versailles
  - Research Site, Verson
  - Research Site, Vert-Saint-Denis
  - Research Site, Verton
  - Research Site, Vertus
  - Research Site, Vervins
  - Research Site, Vestric-et-Candiac
  - Research Site, Vezins
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vénissieux
  - Research Site, Véron
  - Research Site, Vichy
  - Research Site, Vienne
  - Research Site, Vieux-Charmont
  - Research Site, Vieux-Condé
  - Research Site, Vif
  - Research Site, Villard-Bonnot
  - Research Site, Villaudric
  - Research Site, Villebernier
  - Research Site, Villebon-sur-Yvette
  - Research Site, Villebrumier
  - Research Site, Villefagnan
  - Research Site, Villefranche de ROUE
  - Research Site, Villefranche DU PERI
  - Research Site, Villefranche-sur-Mer
  - Research Site, Villefranque
  - Research Site, Villejuif
  - Research Site, Villelongue de LA SA
  - Research Site, Villemoisson SUR ORG
  - Research Site, Villenave-d'Ornon
  - Research Site, Villeneuve LES Mague
  - Research Site, Villeneuve Saint George
  - Research Site, Villeneuve-le-Comte
  - Research Site, Villeneuve-sur-Lot
  - Research Site, Villepinte
  - Research Site, Villepreux
  - Research Site, Villers-Bretonneux
  - Research Site, Villers-Cotterêts
  - Research Site, Villers-Écalles
  - Research Site, Villers-le-Lac
  - Research Site, Villers-Semeuse
  - Research Site, Villersexel
  - Research Site, Villerupt
  - Research Site, Villeurbanne
  - Research Site, Villiers-le-Bel
  - Research Site, Villiers-sur-Marne
  - Research Site, Vincennes
  - Research Site, Viry-Châtillon
  - Research Site, Vitré
  - Research Site, Vitry-le-François
  - Research Site, Vitry-sur-Orne
  - Research Site, Vitry-sur-Seine
  - Research Site, Vitteaux
  - Research Site, Vittel
  - Research Site, Voiron
  - Research Site, Vonnas
  - Research Site, Voujeaucourt
  - Research Site, Vourey
  - Research Site, Walincourt-Selvigny
  - Research Site, Wambrechies
  - Research Site, Wargnies-le-Grand
  - Research Site, Warloy-Baillon
  - Research Site, Warlus
  - Research Site, Warmeriville
  - Research Site, Wasquehal
  - Research Site, Wattignies
  - Research Site, Wattrelos
  - Research Site, Waziers
  - Research Site, Weitbruch
  - Research Site, Weyersheim
  - Research Site, Wingen-sur-Moder
  - Research Site, Wisches
  - Research Site, Yerville
  - Research Site, Yutz
  - Research Site, Yvré-l'Évêque